CLINICAL TRIAL: NCT01093105
Title: A Multicenter, Prospective, Longitudinal, Observational Study of Pediatric Subjects With Globoid Cell Leukodystrophy (Krabbe Disease)
Brief Title: An Observational Study of Pediatric Subjects With Globoid Cell Leukodystrophy (GLD)
Status: Withdrawn | Type: Observational
Why Stopped: Study halted prior to enrollment of first participant
Sponsor: Shire (Industry)
Collaborators: PharmaNet (Industry); Nextrials, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: HGT-GLD-056
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Leukodystrophy, Globoid Cell
Keywords: Leukodystrophy, Globoid Cell; Classic Globoid Cell Leukodystrophy; Early-Onset Globoid Cell Leukodystrophy; Globoid Cell Leukodystrophy; Globoid Cell Leukoencephalopathy; Infantile Globoid Cell Leukodystrophy; Late-Onset Globoid Cell Leukodystrophy; Leukodystrophy, Globoid Cell, Classic; Leukodystrophy, Globoid Cell, Early-Onset; Leukodystrophy, Globoid Cell, Infantile; Leukodystrophy, Globoid Cell, Late-Onset; Psychosine; galactosylsphingosine (psychosine) beta-galactosidase; Psychosine-UDP galactosyltransferase; Krabbe Disease; Krabbe Leukodystrophy; Krabbe's Disease; Krabbe's Leukodystrophy
MeSH Terms: conditions — Leukodystrophy, Globoid Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the natural history of disease progression in infants with globoid cell leukodystrophy (GLD).

DETAILED DESCRIPTION:
This study is being conducted to gather prospective data on disease progression in infants diagnosed with GLD. This study will be performed using protocol-defined, standardized assessments including clinical, developmental, and neurologic measures. All study visits will be conducted in the subject's home. No travel to the study site is necessary.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be considered eligible for this study:

1. The subject has a documented diagnosis of GLD as evidenced by GALC enzyme activity or a GALC genotype that is predictive of GLD.
2. The subject must have clinical signs and symptoms consistent with the diagnosis of infantile GLD including at least 2 of the following:

   1. Chronic difficulty with feeding or unexplained irritability or "fisting" or other signs of abnormal increased tone
   2. CT or MRI imaging, if performed during diagnostic evaluation prior to enrollment, consistent with GLD
   3. Failure to meet at least 2 age-specific developmental milestones consistent with GLD
   4. Loss of deep tendon reflexes or abnormal visual fixation or optic atrophy
3. The subject has documented onset of signs and symptoms consistent with GLD at <12 months of age and is <21 months of age at time of study entry.
4. The subject was born at a gestational age of 35-41 weeks.
5. The subject had a birth weight of ≥2 kg.
6. At study entry, the subject must be able to maintain oral nutrition and hydration without the use of supportive measures, defined as use of a feeding tube.
7. At study entry, the subject must be able to maintain ventilation without the use of invasive supportive measures, defined as use of a breathing tube.
8. The subject must be able, in the opinion of the Investigator, to accommodate the protocol requirements, including feasibility of study visits.
9. The subject's parent(s) or legal guardian must have voluntarily signed an Institutional Review Board/Independent Ethics Committee-approved informed consent form after all relevant aspects of the study have been explained and discussed with the subject's parent(s), or legal guardian.

Exclusion Criteria: Subjects who meet any of the following criteria are not eligible for this study:

1. The subject has neurologic, hearing or vision impairment, difficulty swallowing or feeding, respiratory complications, behavioral disturbances, or other medical conditions that are not due to GLD and are likely to confound the scientific integrity or interpretation of study assessments, as determined by the Investigator.
2. The subject has received treatment with any investigational drug or a device within the 30 days prior to study enrollment through study completion.
3. The subject has received a cord blood or bone marrow transplant or is planning to receive one during the study.
4. The subject's parent(s) or legal guardian is unable to understand the nature, scope, and possible consequences of the study, or does not agree to comply with the protocol defined schedule of assessments.

Max Age: 21 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects with a documented diagnosis of GLD and clinical signs and symptoms consistent with that diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-04-01 (Estimated); Primary Completion 2012-05-01 (Estimated); Study Completion 2012-05-01 (Estimated)

PRIMARY OUTCOMES:
To measure the change from baseline in growth parameters (eg, weight gain, linear growth, head circumference). | 1 year
To determine the onset date of inadequate oral nutrition, hydration, and/or ventilation as a biomarker for survival | 1 year

SECONDARY OUTCOMES:
To assess the change from baseline in clinical parameters of GLD disease progression from a standardized infant neurological examination and infant distress scales. | 1 year
To assess the change from baseline in clinical parameters described in Hagberg's clinical staging. | 1 year
To measure the time to absolute survival | 1 year
To assess the AE experience in this patient population | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda